CLINICAL TRIAL: NCT02511366
Title: The Effect of Repetitive Ileal Brake Activation on Food Intake, Satiety, Gastrointestinal Peptide Release, Gastric Emptying and Gallbladder Volume
Brief Title: Repetitive Brake Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NL50301.068.14
Record Dates: First submitted 2015-04-09; First posted 2015-07-30 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-07

CONDITIONS: Eating; Obesity; Ileal Brake
Keywords: ileal brake
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ileal infusion of casein (Experimental): Ileal infusion of casein
  Interventions: Other: Ileal infusion of casein
- ileal infusion of tap water (Placebo Comparator): ileal infusion of tap water
  Interventions: Other: Ileal infusion of tap water

INTERVENTIONS:
Other: Ileal infusion of casein — Intraileal infusion of casein
  Arms: ileal infusion of casein
Other: Ileal infusion of tap water — Intraileal infusion of tap water
  Other Names: placebo
  Arms: ileal infusion of tap water

SUMMARY:
The appearance of intact macronutrients in the small intestine induces an intestinal brake; a negative feedback mechanism from different parts of the intestine to the stomach, the small intestine and to the central nervous system. These processes inhibit food processing, appetite sensations and food intake, and furthermore they increase feelings of satiety and satiation. Several studies showed that intraileal infusion of nutrients resulted in a reduction in food intake. However only acute effects were investigated in these studies and thus far it is not known whether repetitive (intermittent) infusion results in adaptation to repeated exposure and, thus, a lowered ileal brake response.

ELIGIBILITY:
Inclusion Criteria:

* Based on medical history and previous examination, no gastrointestinal complaints can be defined.
* Age between 18 and 65 years. A higher age comes with a higher chance of comorbidities. These could influence our study outcomes and therefore this age range was chosen. Furthermore, we think this study would be too invasive for subjects over the age of 65. This study will include healthy adult subjects (male and female). Women must be taking contraceptives.
* BMI between 18 and 25 kg/m2)
* Weight stable over at least the last 6 months (≤5% weight change)

Exclusion Criteria:

* History of severe cardiovascular, respiratory, urogenital, gastrointestinal/ hepatic, hematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological/psychiatric diseases, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol. The severity of the disease (major interference with the execution of the experiment or potential influence on the study outcomes) will be decided by the principal investigator.
* Use of medication, including vitamin supplementation, except oral contraceptives, within 14 days prior to testing
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 180 days prior to the study
* Major abdominal surgery interfering with gastrointestinal function (uncomplicated appendectomy, cholecystectomy and hysterectomy allowed, and other surgery upon judgement of the principle investigator)
* Dieting (medically prescribed, vegetarian, diabetic, macrobiological, biological dynamic)
* Pregnancy, lactation
* Excessive alcohol consumption (>20 alcoholic consumptions per week)
* Smoking
* Blood donation within 3 months before the study period
* Self-admitted HIV-positive state
* Evidence of casein or hypersensitivity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Ad libitum food intake | 1 Day
  Ad libitum food intake will be measured in kcal and the end of each test day (4 in total, all within one week)

SECONDARY OUTCOMES:
Satiety | 1 Day
  Visual analogue scale forms for satiety (0-100 mm scale) wil be filled in during each test day (4 in total, all within one week)
Gastrointestinal peptide release (CCK) | 1 Day
  Blood will be drawn during each test day (multiple time points) (4 in total, all within one week)
Gastrointestinal peptide release (GLP-1) | 1 Day
  Blood will be drawn during each test day (multiple time points) (4 in total, all within one week)
Gastrointestinal peptide release (PYY) | 1 Day
  Blood will be drawn during each test day (multiple time points) (4 in total, all within one week)
Gastrointestinal peptide release (insulin) | 1 Day
  Blood will be drawn during each test day (multiple time points) (4 in total, all within one week)
Gastrointestinal peptide release (glucose) | 1 Day
  Blood will be drawn during each test day (multiple time points) (4 in total, all within one week)
gastric emptying rate | 1 Day
  Gastric emptying rate with 13C octanoic acid breath test to determine T1/2
Gallbladder volume | 1 Day
  Gallbladder measurements with ultrasound (volume of GB in mL will be scored)
Small intestinal transit time | 1 Day
  Small intestinal transit time measurements with H2 breath analyser and lactulose

CONTACTS AND LOCATIONS:
Overall Officials: A. Masclee, Prof dr., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Maastricht, Netherlands